CLINICAL TRIAL: NCT01381978
Title: Baseline Study. Obesity Childhood in Cuenca-Ecuador: Prevalence and Risk Factors
Brief Title: Obesity Childhood in Cuenca-Ecuador: Prevalence and Risk Factors
Status: Completed | Type: Observational
Sponsor: Universidad de Cuenca (Other)
Collaborators: University Rovira i Virgili (Other); Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Victoria Abril, MSc Victoria Abril. Researcher University of Cuenca, Universidad de Cuenca
Other Study IDs: DIUC
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Obesity
Keywords: Nutritional status of scholars; Risk factors of obesity; Socioeconomical status; Physical activity habits
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
Hypothesis: Obesity in children of Cuenca is related with socioeconomical status and physical activity habits.

Summary:

The prevalence of obesity and overweigh in all age groups are increasing rapidly in the world. Some factors like physical activity, socioeconomical status, dietary habits, gender, besides genetic factors influence in the development of obesity.

In Cuenca - Ecuador lack information related to prevalence of overweight and obesity in children and the risk factors related.

Socioeconomical status and quality of physical activity are assessed using specially designed questionnaires in a randomized sample of children 6 to 9 years of age of Cuenca city. Nutritional status is assessed using body mass index, relation weight/age and height/age. These data are helpful to develop programs focused to improve nutritional status in scholars of Cuenca.

ELIGIBILITY:
Inclusion Criteria:

* All children of selected sample with an approved consent by their parents

Exclusion Criteria:

* Children with malformations that not permit take anthropometric measures.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children (girls and boys) 6 to 9 years of age. Sample ramdomized of urban schools of Cuenca Ecuador
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2010-10

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Cuenca, Cuenca, Azuay, Ecuador